CLINICAL TRIAL: NCT06825910
Title: Laryngeal Mask Airway I-Gel and Laryngeal Mask Airway Protector for Minor Urological Procedures Under General Anesthesia in Adult Patients: A Randomized Comparative Study
Brief Title: LMA I-Gel Versus LMA Protector During Minor Urological Procedures Under General Anesthesia in Adult Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nikolopoulou Maria Zozefin (Other)
Responsible Party: Sponsor-Investigator, Nikolopoulou Maria Zozefin, Anesthesiology Resident at Sismanoglio General Hospital, Sismanoglio General Hospital
Organization: Sismanoglio General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 19242/29.08.24
Record Dates: First submitted 2025-01-12; First posted 2025-02-13 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-01

CONDITIONS: Airway Management; General Anesthesia
Keywords: LMA; Protector; Airway Device Evaluation; iGel; Airway Device Comparison

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LMA igel group (Active Comparator)
  Interventions: Device: LMA igel
- LMA protector group (Active Comparator)
  Interventions: Device: LMA protector

INTERVENTIONS:
Device: LMA igel — adults allocated to the LMA igel group, an LMA igel device will be inserted intraoperatively
  Arms: LMA igel group
Device: LMA protector — adults allocated to the LMA protector group, an LMA protector device will be inserted intraoperatively
  Arms: LMA protector group

SUMMARY:
This will be a randomized comparative study comparing the two supraglottic devices i-gel and Protector, intraoperatively, during minor urological procedures under general anesthesia in adult patient.

DETAILED DESCRIPTION:
This randomized comparative study aims to evaluate the effectiveness, safety, and unwanted effects of two laryngeal mask airway devices, the iGel and the Protector. The study will involve adult patients during minor urological procedures under general anesthesia. Participants will be divided into two groups: in one group will be inserted the iGel laryngeal mask airway, while in the other group will be inserted the Protector laryngeal mask airway.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II
* Patients older than 18 years
* Procedures in supine and lithotomy position

Exclusion Criteria:

* Tumors or anatomical anomalies of the upper airway
* Known history of difficult intubation
* Limited mouth opening less than 2cm
* Decreased compliance of the lungs or the thoracic cage
* Need of mechanical ventilation after the surgery

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the airway sealing pressure of the Laryngeal Mask Airway (LMA) in neutral, extended, and extended-rotated head positions | Leak pressure will be measured in cmH2O within 60 seconds after successful placement: first in the neutral position, second in the extended position, and third in the extended rotated head position
  After the closure of the adjustable pressure limiting valve (APL) of the ventilation machine with a continuous fresh gas flow of 3L/min, a stethoscope for auscultation will be placed to the lateral position of the thyroid cartilage. Leak pressure is defined as the maximum airway pressure (Ppeak) during which no audible sound, like leak, is detected with the placement of the stethoscope at the thyroid cartilage. Successful placement of the laryngeal mask, will be confirmed right after insertion by the auscultation of both hemithoraces, the indication of capnography, and the ratio of inhaled to exhaled pulmonary volume

SECONDARY OUTCOMES:
Success rate of each device for patients with a potential difficult airway according to the Simplified Airway Index | The patients airway will be evaluated 24 hours before surgery based on the Simplified Airway Index for a potential difficult intubation
  The Simplified Airway Risk Index is a multivariate risk score, ranging from 0 to 12 points, thought to estimate the risk of difficult tracheal intubation based on seven parameters. These seven parameters include the mouth opening, where a mouth opening greater than 4 centimeters between the incisors results in 0 points whereas a distance below results in 1 point, the thyromental distance where thyromental distance greater than 6.5 centimeters results in 0 point whereas a distance between 6-6.5 centimeters is given 1 point and finally a distance below 6 centimeters is given 2 points, the mallampati score where Class I and II of the modified mallampati scoring results in 0 points whereas a class III is given 1 point and a class IV 2 points, the movement of the neck where the ability to move the neck more than 90 degrees results in 0 points whereas a movement range of 80-90 degrees results in 1 point and a movement range below 80 degrees results in 2 points, the ability to underbite mean
The time required for successful placement of the device | Measured from the moment the clinician picks up the LMA device after induction of general anesthesia until the appearance of the first capnography waveform on the monitor with a maximum duration of 60 seconds per attempt and up to three attempts allowed
  This process will involve a maximum of three attempts
Number of attempts to successfully place a nasogastric tube through the specially designed channels of the laryngeal mask | Each attempt, from the moment the clinician picks up the nasogastric tube, will have a time frame of 5 seconds. If the nasogastric tube is not placed within 5 seconds, the attempt will be considered a failure
  The ease of placement will be assessed by counting the number of attempts required to successfully place the nasogastric tube. Success is defined as the ability to place the tube without complications. "Easy" is defined as successful placement on the first attempt, "moderate" as placement on the second attempt, and "difficult" as placement on the third attempt. If placement is not achieved within three attempts, the procedure will be considered unsuccessful.
  Successful placement will by assessed by the successful suction of gastric fluid
Documentation of adverse events after the exertion | Immediately after the exertion
  Complications like blood-stain visible on the LMA after exertion and post-operative sore throat

CONTACTS AND LOCATIONS:
Locations (1):
- SismanoglioGH, Athens, Greece

IPD SHARING:
Plan to Share IPD: No